CLINICAL TRIAL: NCT01227746
Title: A Retrospective Study of C-kit Mutation Status in Asian Patients With Advanced Gastro-intestinal Stromal Tumors (GIST) Treated With Imatinib.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: GA03/17/10
Record Dates: First submitted 2010-10-21; First posted 2010-10-25 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Asian Patients With Advanced Gastro-intestinal Stromal Tumors (GIST) Treated With Imatinib
Keywords: Advanced gastro-intestinal stromal tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tumor biopsies
  Interventions: Procedure: Tumor biopsies

INTERVENTIONS:
Procedure: Tumor biopsies

SUMMARY:
Imatinib is the current standard treatment for advanced GIST. Previous studies have shown that GIST genotype was associated with treatment outcomes with exon 11 having superior outcome compared with exon 9 or WT.10, 11 In patients with exon 9 kit mutation, the response rate was higher at when imatinib was given at 800mg daily compared with the standard dose of 400mg daily. Although the data linking tyrosine kinase mutation status and imatinib response in metastatic GISTs is intriguing, more information is needed before mutation testing is adopted as part of the routine analysis of high-risk or overtly malignant KIT-expressing GISTs.25 Despite the fact that exon 9 mutations are associated with a lower response rate, overall survival does not appear to be better with high-dose therapy. The investigators propose to conduct a retrospective analysis of mutational analysis on patients with GIST and determine the relationship between patient response and imatinib dose.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of advanced stage or metastatic GIST
2. Asian patient (as defined by the investigator)
3. First line treatment with imatinib
4. Availability of tumor samples for kit mutation analysis
5. Availability of tumor response rate and or time to progression data

Exclusion Criteria:

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asian patients with advanced gastro-intestinal stromal tumors (GIST) treated with imatinib.
Sampling Method: Non-Probability Sample
Dates: Start 2011-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Tornillo L, Terracciano LM. An update on molecular genetics of gastrointestinal stromal tumours. J Clin Pathol. 2006 Jun;59(6):557-63. doi: 10.1136/jcp.2005.031112. PMID 16731599
- [Background] Heinrich MC, Corless CL, Duensing A, McGreevey L, Chen CJ, Joseph N, Singer S, Griffith DJ, Haley A, Town A, Demetri GD, Fletcher CD, Fletcher JA. PDGFRA activating mutations in gastrointestinal stromal tumors. Science. 2003 Jan 31;299(5607):708-10. doi: 10.1126/science.1079666. Epub 2003 Jan 9. PMID 12522257